CLINICAL TRIAL: NCT06841432
Title: Endoscopic Coblation Versus Suction Diathermy in Pediatric Adenoidectomy: Randomized Clinical Trial
Brief Title: Coblation Versus Suction Diathermy in Pediatric Adenoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Nabil Selim, Resident doctor of otorhinolanrgology at alazhar univeristy hopsital in assiut, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSCAZASTENT03028
Record Dates: First submitted 2025-02-06; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adenoid Hypertrophy; Adenoidectomy; Coblation Adenoidectomy; Suction Daithermy
Keywords: Endoscopic; Adenoidectomy; adenoid hypertrophy; Pediatric; Suction Diathermy; Coblation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients who underwent the adenoidectomy using suction diathermy (Active Comparator): One hundred and five patients underwent a suction diathermy adenoidectomy procedure. The soft palate was gently retracted using two suction catheters, allowing a 70-degree angled endoscope (Storz, Germany) placed in the oropharynx to provide a clear view of the adenoidal tissue and surrounding structures in the nasopharynx. Using a malleable size 10 or 12 French hand-switching suction coagulator, the adenoidal tissue was carefully ablated, starting from the uppermost part. The procedure was completed when the posterior choanae were clearly visible, and the nasopharynx had a smooth, unobstructed appearance. Great care was taken to avoid injuring the Eustachian tube orifice, posterior septum, choanae, inferior turbinate, palate, and posterior pharyngeal wall. Continuous irrigation with saline, either through the mouth or the nose, helped minimize any thermal damage caused by the diathermy machine.
  Interventions: Procedure: adenoidectomy by Suction diathermy
- patients who underwent the adenoidectomy using coblation (Experimental): One hundred and five patients underwent a Coblation-assisted adenoidectomy procedure. The child was positioned in Rose's position, which helped retract the soft palate and improve visibility of the nasopharynx. Two soft rubber catheters were inserted into the patient's mouth, with the distal and proximal ends crossed externally and secured with a clamp. The COBLATOR™ II surgery system Model EC8000-01 was used, with a power setting of nine for ablation and five for coagulation. Under general anesthesia, the adenoidectomy was performed using either a 4 mm, 70-degree angled endoscope inserted orally or a zero-degree endoscope inserted through the nose, providing effective visualization of the nasopharynx. After the procedure, hemostasis was achieved by using a combination of the coagulation and ablation modes.
  Interventions: Procedure: adenoidectomy using coblatioion

INTERVENTIONS:
Procedure: adenoidectomy using coblatioion — One hundred and five patients underwent a Coblation-assisted adenoidectomy procedure. The child was positioned in Rose's position, which helped retract the soft palate and improve visibility of the nasopharynx. Two soft rubber catheters were inserted into the patient's mouth, with the distal and proximal ends crossed externally and secured with a clamp. The COBLATOR™ II surgery system Model EC8000-01 was used, with a power setting of nine for ablation and five for coagulation. Under general anesthesia, the adenoidectomy was performed using either a 4 mm, 70-degree angled endoscope inserted orally or a zero-degree endoscope inserted through the nose, providing effective visualization of the nasopharynx. After the procedure, hemostasis was achieved by using a combination of the coagulation and ablation modes.
  Arms: patients who underwent the adenoidectomy using coblation
Procedure: adenoidectomy by Suction diathermy — One hundred and five patients underwent a suction diathermy adenoidectomy procedure. The soft palate was gently retracted using two suction catheters, allowing a 70-degree angled endoscope (Storz, Germany) placed in the oropharynx to provide a clear view of the adenoidal tissue and surrounding structures in the nasopharynx. Using a malleable size 10 or 12 French hand-switching suction coagulator, the adenoidal tissue was carefully ablated, starting from the uppermost part. The procedure was completed when the posterior choanae were clearly visible, and the nasopharynx had a smooth, unobstructed appearance. Great care was taken to avoid injuring the Eustachian tube orifice, posterior septum, choanae, inferior turbinate, palate, and posterior pharyngeal wall. Continuous irrigation with saline, either through the mouth or the nose, helped minimize any thermal damage caused by the diathermy machine.
  Arms: patients who underwent the adenoidectomy using suction diathermy

SUMMARY:
The goal of this clinical trial is to compare two surgical procedures in endoscopic adenoidectomy including Coblation and Suction diathermy

. The main questions it aims to answer are: Does the Coblation device have less time, less pain, less postoperative crustation and bad odor, less intraoperative bleeding, and less recurrence?

Participants will:

will undergo both procedures every day for 6 months Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* all patients aged 2 to 18 years
* patients who had isolated adenoid hypertrophy
* patients' hemoglobin levels above 10 mg/dl

Exclusion Criteria:

* those with recent upper respiratory tract infections, evidence of bleeding disorders, serous otitis media, chronic tonsillitis
* those advised against undergoing adenoidectomy after consulting a phoniatrist
* patients with atrophic rhinitis those with nasal obstruction caused by other nasal or paranasal conditions such as inferior turbinate hypertrophy, Choanal atresia, deviated nasal septum, antrochoanal polyps, and other causes of nasal obstruction in children.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Operative duration | During the procedure
  The procedure, from the initial insertion of the Bowel-Davis mouth gag to the complete removal of the adenoid and the gag, was timed in minutes.
Intraopertive blood loss | during the procedures
  Boezaart surgical field grading scale was used to evaluate the intraoperative bleeding
Postopertaive Pain | Patients reported their pain levels every day before taking any pain medication during the 7 days after their surgery
  The Wong-Baker Pain Scale consists of 6 faces depicting different levels of pain. Face 1 represents no pain, Face 2 indicates a little bit of hurt, Face 3 indicates a little more hurt, Face 4 indicates even more hurt, Face 5 indicates a whole lot of hurt, and Face 6 indicates the worst possible hurt, with pain scores ranging from 0 to 10. Both the children and their parents were informed about the purpose of the questionnaires and how to fill them out before the surgery

SECONDARY OUTCOMES:
Development of bad breath | from the end of operation till 2 weeks post operation
  frequency of Children who presented with bad breath
recovery time | three months post opertaive
  time which was talken for the patients to resume their normal social routines
secondary bleeding | up to one month surgery
  frequency of Children who presented with bleeding that occurred after 24 hrs of operation
Pre- and post-adenoid size grading | preintervention (one day before opertaion ) and postintervention (up to three months)
  The Parikh grading system (1-4) is used to assess the extent of adenoid tissue contact with surrounding structures: Grade 1 - adenoid tissue not in contact, Grade 2 - adenoid tissue in contact with Eustachian tube cushions, Grade 3 - adenoid tissue in contact with vomer, Grade 4 - adenoid tissue in contact with soft palate

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar university Hopital in Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided